CLINICAL TRIAL: NCT00290212
Title: Phase II Study of Natto Supplementation to Prevent Loss of Bone Mass in Women Immediately After Menopause: a Randomised Double Blind Placebo-Controlled Trial
Brief Title: Natto Supplementation to Prevent Loss of Bone Mass in Women Immediately After Menopause
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other); The International Osteoporosis Foundation (Other); Haukeland University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REK V 77/2005
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2006-12

CONDITIONS: Perimenopausal Bone Loss
Keywords: Women; Bone density; Menopause; Dietary Supplements; Vitamin K2
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Soy Foods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Natto capsules (food suppl.) cont. 360 microg. vit K2/day
Drug: Placebo capsules

SUMMARY:
Study Objective: To determine whether Natto supplementation in women immediately after menopause might prevent severe bone loss

Study population: Women 50 - 60 years, 1-5 years after menopause

Study Design: Double-blind, placebo-controlled, randomized controlled trial. A "phase II" clinical trial.

Instruments Used to Measure Therapeutic Response: Lunar Prodigy DEXA bone densitometer

Study Treatment Group: Daily supplementation with Vitamin K2, "NATTO"

Study Control Group: Identically-looking placebo medication

Duration of treatment: 12 months

Duration of Subject Participation in Study: 12 months Assessment of Therapeutic response: Given an expected reduction of bone mass density of - 1.1% annually in the placebo group, the minimum clinically significant difference between the groups is 0.3 percentage points. The trial is therefore powered to detect a reduction in annual bone mass loss of 0.3 percentage points in the treatment group.

Numbers of Evaluable Subjects Required: 304 Maximum # Subjects 334

ELIGIBILITY:
Inclusion Criteria:

* Women living in the city of Tromsø, not using hormone replacement therapy, 1-5 years after menopause.

Exclusion Criteria:

* History of hip fracture
* Bone disease affecting bone mineral density
* Use of vitamin K antagonists
* Significant co-morbidity that makes it difficult to obtain BMD measurements
* Use of hormone replacement therapy or other therapy that influence bone remodeling

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 304 (Actual)
Dates: Start 2006-01; Study Completion 2007-06

PRIMARY OUTCOMES:
Bone mass density

CONTACTS AND LOCATIONS:
Overall Officials: Nina Emaus, MSc PhD, Principal Investigator — NAFKAM, Fac.of Medicine, Univ. of Tromsø, Norway; Sameline Grimsgaard, MD, MPH, PhD, Principal Investigator — University Hospital of North Norway; Vinjar Fønnebø, MD, MSc, PhD, Study Chair — NAFKAM, University of Tromsø, Norway
Locations (2):
- Norway (2):
  - Clinical Research Center, University Hospital of North Norway, Tromsø, Tromsø
  - Haukeland University Hospital, Bergen